CLINICAL TRIAL: NCT04208503
Title: Ultrasound and Functional Thyroid Evaluation in Preterm Infants Born Between 24 and 32 Weeks of Gestation
Brief Title: Ultrasound and Functional Thyroid Evaluation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Princess Anna Mazowiecka Hospital, Warsaw, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: 3/2019
Record Dates: First submitted 2019-12-13; First posted 2019-12-23 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Thyroid; Gland; Functional Disturbance
Keywords: thyroid volume; ultrasound; preterm infants; thyroid hormone
MeSH Terms: conditions — Thyroid Diseases | interventions — Diagnostic Tests, Routine; Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — 1 ml blood for TSH and FT4 assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: thyroid ultrasound — After meeting enrolment criteria the thyroid ultrasound will be performed at 32 and 36 weeks of gestation, blood test for TSH and FT4 will be obtained at 14-21 day of life, at 32 and 36 weeks of gestation
  Other Names: Diagnostic test; blood test for TSH and FT4 concentration

SUMMARY:
Thyroid disorders are most commonly concomitant with prematurity and still remains a controversial topic. The incidence of a temporary form of hypothyroidism among preterm neonates is higher than in the general population. Transient prematurity hypothyroxinemia is defined as a temporary reduction in FT4 values without increase in TSH values. Currently, there is no consensus about normal thyrotropine (TSH) and free thyroxine (FT4) values in preterm infants.

The aim of this study is to determine the volume of the thyroid gland in preterm infants born between 24 and 32 weeks of gestation inborn or admitted to the unit within 14 days from birth and compare it with the results of TSH and FT4 blood concentration. Besides, the objective of the study is to determine values of thyroid hormones in premature infants born before 33 wk gestation to help neonatologist to interpreter the thyroid hormone results

DETAILED DESCRIPTION:
Thyroid disorders are most commonly concomitant with prematurity and still remains a controversial topic. Preterm infants are susceptible to thyroid disorders due to many reasons including immaturity of hypothalamopituitary-thyroid axis, non-thyroidal illness, impaired synthesis and metabolism of thyroid hormones, medication administration like dopamine, steroids, caffeine.The incidence of a temporary form of hypothyroidism among preterm neonates is higher than in the general population. Transient prematurity hypothyroxinemia is defined as a temporary reduction in FT4 values without increase in TSH values. It is a diagnostic challenge in order to differentiate it from thyroid disfunction in the critically ill patient. Currently, there is no consensus about normal thyrotropine (TSH) and free thyroxine (FT4) values in preterm infants. Given the delayed appearance of TSH value increase in preterm newborns additional thyroid evaluation methods are sought. We believe the thyroid ultrasound might prove helpful.

The aim of this study is to determine the volume of the thyroid gland in preterm infants born between 24 and 32 weeks of gestation inborn or admitted to the unit within 14 days from birth and compare it with the results of TSH and FT4 blood concentration. We will performed the thyroid ultrasound to estimate the thyroid volume to aid in the comparative evaluation of infants with suspected thyroid disease. The value of sonography thyroid volume will give specialists possibility to identify a gland as normal, small or enlarged. Besides, the objective of the study is to determine value of thyroid hormones in premature infants born before 33 wk gestation to help neonatologist to interpreter the thyroid hormone results

ELIGIBILITY:
Inclusion Criteria:

* preterm infants born between 24 and 32 weeks of gestation (estimated by ultrasound)
* in born or admitted to the unit within one week from birth
* randomization within 7 days from birth
* parental consent

Exclusion Criteria:

* preterm delivery <23 weeks of gestation or > 32 weeks (estimated by ultrasound)
* major congenital abnormalities
* no parental consent
* medications used after birth: steroids, vasopressors (up to 12 hours after end of treatment)
* positive thyroid stimulating antibodies (TSAb) in the mother
* mothers with thyroid disease treated with antythyroid drugs
* mothers treated with amiodarone

Ages: 1 Week to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We plan to recruit all consecutive preterm infants born ≤ 32 weeks of gestation.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Determination of FT4 and TSH values in preterm infants born at 24-28 weeks of gestation | 14-21 days of life, at 32 and 36 weeks of PCA
  FT4 and TSH - blood concentration
Determination of FT4 and TSH values in preterm infants born at 29-32 weeks of gestation | at 14-21 day of life, at 32 and 36 weeks of PCA
  FT4 and TSH - blood concentration
Determination of ultrasound thyroid volume in both groups of preterm infants (i.e., those born at 24-28 weeks of gestation and those born at 29-32 weeks of gestation) | at 32 and 36 weeks of PCA
  The thyroid volume
Evaluation of correlations between circulating thyroid hormone concentrations and thyroid volume | at 32 and 36 weeks of PCA
  comparison of values of FT4, TSH and thyroid volume

SECONDARY OUTCOMES:
Comparison of changes in FT4 evaluated at 32 and 36 weeks of PCA in each group of preterm infants | at 14-21 day of life, at 32 and 36 weeks of PCA
  comparison of results
Comparison of changes in TSH evaluated at 32 and 36 weeks of PCA in each group of preterm infants | 14-21 days of life, at 32 and 36 weeks of PCA
  comparison of results
Analysis of TSH values over time (to determine the optimal time for TSH measurement) | at 14-21 day of life, at 32 and 36 weeks of PCA
  Intervention time
Evaluation of changes in ultrasound thyroid volume examined at 32 and 36 weeks of PCA in each group of preterm infants | at 32 and 36 weeks of PCA
  comparison of results
Evaluation of the correlation between thyroid volume and circulating thyroid hormone concentrations with the head circumference and body mass at 32 and 36 weeks of PCA | at 32 and 36 weeks of PCA
  correlation of results with the body mass and the head circumference

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Mikolajczak, MD PhD, Study Chair — Princess Anna Mazowiecka
Locations (1):
- Department of Neonatology and Neonatal Intensive Care Warsaw Medical University, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be available, after deidentiﬁcation. The study protocol will also be available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2021-December 2021
Access Criteria: Documents will be accessible to anyone who provides a methodologically sound proposal immediately following publication with no end date.

REFERENCES:
- [Background] Chaudhari M, Slaughter JL. Thyroid Function in the Neonatal Intensive Care Unit. Clin Perinatol. 2018 Mar;45(1):19-30. doi: 10.1016/j.clp.2017.10.005. Epub 2017 Dec 13. PMID 29406004
- [Background] McGrath N, Hawkes CP, Mayne P, Murphy NP. Optimal Timing of Repeat Newborn Screening for Congenital Hypothyroidism in Preterm Infants to Detect Delayed Thyroid-Stimulating Hormone Elevation. J Pediatr. 2019 Feb;205:77-82. doi: 10.1016/j.jpeds.2018.09.044. Epub 2018 Oct 24. PMID 30529133
- [Background] Radetti G, Zavallone A, Gentili L, Beck-Peccoz P, Bona G. Foetal and neonatal thyroid disorders. Minerva Pediatr. 2002 Oct;54(5):383-400. English, Italian. PMID 12244277
- [Background] Vigone MC, Caiulo S, Di Frenna M, Ghirardello S, Corbetta C, Mosca F, Weber G. Evolution of thyroid function in preterm infants detected by screening for congenital hypothyroidism. J Pediatr. 2014 Jun;164(6):1296-302. doi: 10.1016/j.jpeds.2013.12.048. Epub 2014 Feb 8. PMID 24518164
- [Background] Khan SS, Hong-McAtee I, Kriss VM, Stevens S, Crawford T, Hanna M, Bada H, Desai N. Thyroid gland volumes in premature infants using serial ultrasounds. J Perinatol. 2018 Oct;38(10):1353-1358. doi: 10.1038/s41372-018-0149-0. Epub 2018 Jul 30. PMID 30061589
- [Background] Oh KW, Koo MS, Park HW, Chung ML, Kim MH, Lim G. Establishing a reference range for triiodothyronine levels in preterm infants. Early Hum Dev. 2014 Oct;90(10):621-4. doi: 10.1016/j.earlhumdev.2014.07.012. Epub 2014 Aug 24. PMID 25150803
- [Background] Kurtoglu S, Ozturk MA, Koklu E, Gunes T, Akcakus M, Yikilmaz A, Buyukkayhan D, Hatipoglu N. Thyroid volumes in newborns of different gestational ages: normative data. Arch Dis Child Fetal Neonatal Ed. 2008 Mar;93(2):F171. doi: 10.1136/adc.2007.130211. No abstract available. PMID 18296580
- [Background] Goldis M, Waldman L, Marginean O, Rosenberg HK, Rapaport R. Thyroid Imaging in Infants. Endocrinol Metab Clin North Am. 2016 Jun;45(2):255-66. doi: 10.1016/j.ecl.2016.02.005. PMID 27241963
- [Background] Knobel RB. Thyroid hormone levels in term and preterm neonates. Neonatal Netw. 2007 Jul-Aug;26(4):253-9. doi: 10.1891/0730-0832.26.4.253. PMID 17710960
- [Background] Kaluarachchi DC, Colaizy TT, Pesce LM, Tansey M, Klein JM. Congenital hypothyroidism with delayed thyroid-stimulating hormone elevation in premature infants born at less than 30 weeks gestation. J Perinatol. 2017 Mar;37(3):277-282. doi: 10.1038/jp.2016.213. Epub 2016 Dec 1. PMID 27906195